CLINICAL TRIAL: NCT05742308
Title: The Effect of Laughter Yoga on Hope and School Burnout Among Secondary School Students: A Parallel Group Randomized Control Trial.
Brief Title: The Effect of Laughter Yoga on Hope and School Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nilgun Kuru Alici, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D6907
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Laughter Therapy; Laughter Yoga; Hope; School Burnout
MeSH Terms: conditions — Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Laughter yoga (Experimental): The intervention group received laughter yoga twice a week for three weeks.
  Interventions: Behavioral: Laughter yoga
- No Intervention: Control group (No Intervention): The control group did not take part in the laughter yoga program.

INTERVENTIONS:
Behavioral: Laughter yoga — Laughter yoga program was composed of four steps. The first step, which took 10 minutes, had warm-up exercises including gentle stretching and hand clapping. The second step, which included deep breathing exercises and hand clapping, took 5 minutes. The third step involved children's games and laughter exercises. The sessions included a combination of different laughter exercises. The last step, which included yoga nidra took 5 minutes.
  Arms: Experimental: Laughter yoga

SUMMARY:
This study aimed to evaluate the effect of laughter yoga on hope and school burnout among secondary school (8th Grade) students. The study hypothesized that laughter yoga would have an effect on hope and school burnout scores among secondary school students

DETAILED DESCRIPTION:
Purpose: The aim of the research was to examine the effects of laughter yoga on life hope and school burnout among secondary school (8th Grade) students.

Methods: The study was conducted with 60 (30 in the intervention group, and 30 in the control group) students. The study population consisted of 8th grade students. Laughter yoga sessions were applied to the intervention group twice a week for 6 weeks. No intervention was offered to the control group. Data were collected by a socio-demographic questionnaire, school burnout inventory and Children's Hope Scale.

Results: After laughter yoga, the intervention result showed a significant decrease in burnout (d=0.129; p < 0.001) and increase hope scores (d=0.556; p < 0.001) compared to the control group.

Conclusion: The study reveals that laughter yoga affects students' burnout and hope levels. It is recommended to organize laughter yoga activities in schools to decrease burnout and increase hope of students.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the study were determined as being an 8th-grade student, speaking and understanding Turkish, and being able to perform daily life activities.

Exclusion Criteria:

* having severe hearing or perceptual deficits that impaired communication; having dementia, Alzheimer's disease, depression, uncontrolled diabetes, hypertensive disease and surgical operations with the risk of bleeding.

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Children's Hope Scale scores | up to 6 weeks
  The Children's Hope Scale (CHS) is self-report measure of children's perceptions that their goals can be met. The CHS consists of six items that are hypothesized to relate to the two underlying factors of agency and pathways. Adding the response values for pathway questions will provide a pathway score ranging from 2-12; higher scores reflect higher pathways thinking. Adding the response values for agency questions will provide an agency score ranging from 2-12; higher scores reflect higher agency thinking. Adding pathway and agency scores will provide an overall hope score (i.e., level of hope). Scores of 4-8 indicate no to very low hope, 9-12 indicate slightly hopeful, 13-16 indicate moderately hopeful, and 17-24 indicates highly hopeful.

SECONDARY OUTCOMES:
School Burnout Inventory score | up to 6 weeks
  Burnout is assessed in accordance with the School Burnout Inventory scale comprises nine uni dimensional items measuring the three dimensions: (1) exhaustion at school (e.g., I feel overwhelmed by my school work; I brood over matters related to my school work a lot during my free time); (2) disengagement or cynicism with regard to the meaning of school (e.g., I feel a lack of motivation in my school work and often think of giving up; I feel that I am losing interest in my school work), and (3) feelings of inadequacy at school (e.g., I often have feelings of inadequacy with regard to my school work). There were three items for each of the three dimensions, all of which were rated on a six-point scale (1 = strongly disagree; 6 = strongly agree). We calculated separate sum scores at each of the four time points for the three dimensions and the overall burnout.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kuru Alici, PhD, Principal Investigator — Associate professor
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuru Alici N, Kalanlar B. Effect of Laughter Yoga on School Burnout and Hope Among Secondary School (Eighth Grade) Students: A Parallel Group Randomized Control Trial. Florence Nightingale J Nurs. 2024 Feb 28;32(1):68-74. doi: 10.5152/FNJN.2024.23200. PMID 39555642